CLINICAL TRIAL: NCT03401918
Title: Assessing the Endometrial Environment in Recurrent Pregnancy Loss and Unexplained Infertility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40761
Record Dates: First submitted 2018-01-01; First posted 2018-01-17 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Pregnancy Loss; Unexplained Infertility
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with recurrent pregnancy loss or unexplained infertility (Experimental): Patients with recurrent pregnancy loss or unexplained infertility will have an assessment of the uterine environment at the time of implantation, followed by testing of uterine endometrial gene expression using the ERA test and the uterine micro biome.
  Those who have abnormal results (an abnormal microbiome or an abnormal ERA) will have the option to undergo treatment followed by retesting of the uterine environment. For an abnormal ERA suggesting a pre-receptive result, luteal phase vaginal progesterone supplementation will be offered prior to re-testing of the ERA. For an abnormal microbiome a combination of oral antibiotics and vaginal probiotics will be offered prior to re-testing the uterine microbiome.
  Interventions: Diagnostic Test: Uterine ERA and microbiome testing; Drug: Oral antibiotics and vaginal probiotics
- Healthy Control Patients (Experimental): Patients who have had a normal delivery and no history of infertility or recurrent pregnancy loss will have assessment of the uterine environment at the time of implantation.
  Interventions: Diagnostic Test: Uterine ERA and microbiome testing

INTERVENTIONS:
Diagnostic Test: Uterine ERA and microbiome testing — Uterine fluid and endometrial biopsy collection to test uterine endometrial receptivity array and microbiome.
Drug: Oral antibiotics and vaginal probiotics — For subjects with abnormal microbiome results, oral antibiotics and vaginal probiotic treatment will be offered followed by a repeat uterine microbiome biopsy.
  Arms: Patients with recurrent pregnancy loss or unexplained infertility

SUMMARY:
The purpose of this study is to determine if patients with recurrent pregnancy loss or unexplained infertility have an altered uterine gene expression or uterine microbiome (micro-organism composition) during the window of embryo implantation. Furthermore we would like to assess for women with an abnormal uterine gene expression whether vaginal progesterone medication improves or alters gene expression and for women with an abnormal microbiome whether antibiotic treatment followed by probiotic treatment normalizes the microbiome.

DETAILED DESCRIPTION:
Recurrent pregnancy loss and unexplained infertility are emotional and difficult diagnoses. Despite a thorough medical investigation, many cases of recurrent pregnancy loss and infertility remain unexplained. Understanding endometrial factors that may contribute to these diseases may lead to improved treatment options in the future. The purpose of this study is to determine if patients with recurrent pregnancy loss or unexplained infertility have an altered uterine gene expression or uterine microbiome (micro-organism composition) during the window of embryo implantation. Furthermore we would like to assess for women with an abnormal uterine gene expression whether vaginal progesterone medication improves or alters gene expression and for women with an abnormal microbiome whether antibiotic treatment followed by probiotic treatment normalizes the microbiome.

A standard evaluation for infertility includes a uterine cavity evaluation, evaluation for ovarian reserve testing, and for patients with recurrent pregnancy loss parental testing for uterine infection, chromosome analysis, autoimmune and thyroid screening. This standard workup, however, does not include a molecular or microbial assessment of the endometrium. Endometrial factors may contribute to unexplained infertility or recurrent pregnancy loss however the extent of this is unknown.

We are recruiting patients who have recurrent pregnancy loss, unexplained infertility, and healthy control patients who have had a term delivery in order to compare differences between these groups.

Subjects will undergo an endometrial biopsy that will specifically test the receptivity of your endometrium as well as identify the bacterial composition of the uterine environment (microbiome). The endometrial receptivity array and microbiome testing will be performed at no cost. The endometrial receptivity array provides information on the receptivity of a patient's endometrium to the implantation of an embryo. This may yield additional information regarding the etiology of a patient's infertility and/or recurrent pregnancy loss. If this testing is abnormal we may repeat the biopsy after vaginal progesterone supplementation to see if this normalizes the results. If the microbiome is abnormal we may repeat the biopsy after oral antibiotics and vaginal probiotics to see if this normalizes your microbiome results.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

1. Recurrent Pregnancy Loss

   Inclusion:
   * Age 18-45
   * 3 or more SABs including biochemical pregnancies OR 2 or more SABs if one is documented to be euploid

   Exclusion:
   * irregular menstrual cycles
   * Submucosal fibroid >3cm
   * Stage 3-4 endometriosis
   * BMI >40
   * IUD within the last 3 months
2. Unexplained infertility Patients

   Inclusion:
   * TTC x >= 1 year
   * At least one SA with TMS >10 mil within last 2 years
   * At least one patent fallopian tube documented by HSG or SHG
   * Cycle length 25-35 days

   Exclusion:
   * Irregular menstrual cycles
   * Submucosal fibroid >3cm
   * Stage 3-4 endometriosis
   * BMI >40
   * IUD within the last 3 months
   * Less then 2 SABs including biochemical pregnancies
3. Healthy control patients

Inclusion:

* Patients who present for fertility preservation, sex selection, same sex couples needing fertility care, preconception counseling
* 1 or more live births

Exclusion:

* Irregular menstrual cycles
* Submucosal fibroid >3cm
* Stage 3-4 endometriosis
* BMI >40
* IUD within the last 3 months
* Less then 2 SABs including biochemical pregnancies
* No history of RPL or infertility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Endocrinology and Infertility Center at Stanford University, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
Started | 25 | 16
Completed | 25 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients | Total
Number analyzed (Participants) | 25 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 16 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 2 | 15
  Caucasian | 12 | 12 | 24
  Black | 0 | 1 | 1
  Hispanic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Microbiome Bacterial Sequencing
Description: The primary outcome will abnormal microbiome results. An abnormal microbiome will be defined as less then 90% lactobacilli on DNA sequencing
Time Frame: 1 month
Population: No participants were analyzed because the assay failed validation and the results are uninterpretable.
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Abnormal Endometrial Receptivity Array
Description: The second primary outcome will be abnormal endometrial receptivity array defined as non-receptive (pre or post receptive) based on RNA sequencing of an endometrial gene array.
Time Frame: 1 month
Population: No endometrial receptivity array data were collected because the microbiome assay failed validation and further testing was not done.
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Normalized Microbiome Bacterial Sequencing
Description: The primary outcome will be normal microbiome results defined as >90% lactobacilli after oral antibiotics and vaginal probiotics after initially abnormal microbiome results
Time Frame: 3-6 months
Population: Data were not collected for this outcome measure as the study did not continue to the treatment phase.
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Normalized Endometrial Receptivity Array
Description: The primary outcome will be normal endometrial receptivity array results defined as receptive after luteal phase progesterone support after initially abnormal endometrial receptivity array results
Time Frame: 3-6 months
Population: Data were not collected for this outcome measure as the study did not continue to the treatment phase.
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Patients With Recurrent Pregnancy Loss or Unexplained Infertility | Healthy Control Patients
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 0/25 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03401918/Prot_000.pdf
  • Informed Consent Form (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03401918/ICF_001.pdf